CLINICAL TRIAL: NCT07186868
Title: A Prospective, Open-Label, Single-Arm Study of Iparomlimab and Toripalimab Plus Nab-Paclitaxel With or Without Bevacizumab in Recurrent/Metastatic Cervical Cancer Progressed on Anti-PD-(L)1 Therapy
Brief Title: QL706 + Chemo ± Bevacizumab in Anti-PD-(L)1-Resistant R/M Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC-01
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Cervical Cancer; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QL1706 + Nab-Paclitaxel ± Bevacizumab: All participants will receive the study intervention: Iparomlimab and Tuvonralimab (QL1706) at 5.0 mg/kg IV Q3W + Nab-Paclitaxel at 260 mg/m² IV Q3W, with or without Bevacizumab (7.5-15 mg/kg IV Q3W) per investigator's choice, for 6 cycles. This is followed by maintenance therapy with QL1706 ± Bevacizumab until disease progression, unacceptable toxicity, or other discontinuation criteria are met.
  Interventions: Biological: Iparomlimab and Tuvonralimab (QL1706) + Nab-Paclitaxelwith or without Bevacizumab

INTERVENTIONS:
Biological: Iparomlimab and Tuvonralimab (QL1706) + Nab-Paclitaxelwith or without Bevacizumab — All participants will receive the study intervention: Iparomlimab and Tuvonralimab (QL1706) at 5.0 mg/kg IV Q3W + Nab-Paclitaxel at 260 mg/m² IV Q3W, with or without Bevacizumab (7.5-15 mg/kg IV Q3W) per investigator's choice, for 6 cycles. This is followed by maintenance therapy with QL1706 ± Bevacizumab until disease progression, unacceptable toxicity, or other discontinuation criteria are met.

SUMMARY:
This is a clinical research study for women with recurrent or metastatic cervical cancer whose disease has progressed after prior treatment with a PD-1/PD-L1 inhibitor immunotherapy.

The study will evaluate the effectiveness and safety of a new combination treatment consisting of iparvolimab and tuvonralimab (QL1706)-a dual-targeting immunotherapy drug-along with chemotherapy (nab-paclitaxel) with or without bevacizumab, an anti-angiogenic drug that may help prevent tumor growth.

Approximately 25 participants will be enrolled in this open-label, single-arm study. All participants will receive the study treatment for up to 6 cycles, followed by maintenance therapy until disease progression, unacceptable side effects, or other reasons for stopping treatment.

The main goal of the study is to see how many patients respond to the treatment (Objective Response Rate, ORR). Other goals include measuring how long the response lasts, how long patients live without the cancer getting worse, and overall survival. Safety and quality of life will also be closely monitored.

This study is for women aged 18-75 who have previously received PD-1/PD-L1 treatment and whose cancer has worsened. Participants must be in generally good health with adequate organ function and no other active cancers.

The study will be conducted at a single center in China. All participants will provide written informed consent before joining the study.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm, single-center phase II clinical trial investigating the efficacy and safety of a combination therapy in patients with recurrent or metastatic cervical cancer who have experienced disease progression following prior anti-PD-1/PD-L1 therapy.

The study aims to address the high unmet medical need in this patient population where treatment options are limited after failure of immunotherapy. The investigational regimen consists of iparomlimab and tuvonralimab (QL1706), a novel bifunctional antibody targeting both PD-1 and CTLA-4, combined with nab-paclitaxel chemotherapy, with the optional addition of bevacizumab at the investigator's discretion.

Approximately 25 participants will receive the combination treatment for 6 cycles (3-week cycles), followed by maintenance therapy with QL1706 ± bevacizumab until disease progression, unacceptable toxicity, or other discontinuation criteria are met. The primary endpoint is Objective Response Rate (ORR) per RECIST 1.1. Secondary endpoints include Progression-Free Survival (PFS), Duration of Response (DoR), Disease Control Rate (DCR), Overall Survival (OS), and safety profile. An exploratory objective will analyze the correlation between PD-L1 expression status and treatment outcomes.

The study will include rigorous safety monitoring per NCI CTCAE v5.0 guidelines and regular tumor assessments. The sample size was calculated based on the assumption of improving the ORR from a historical control of 15% to 40% with the new combination.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 75 years.
* Histologically, pathologically, or radiologically confirmed recurrent or metastatic cervical cancer.
* At least one measurable lesion as defined by RECIST 1.1 (non-nodal lesion longest diameter ≥10 mm or lymph node short axis ≥15 mm).
* ECOG performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* Disease progression after receiving at least one prior anti-PD-1/PD-L1 monoclonal antibody therapy (alone or in combination).
* Adequate organ function within 14 days before enrollment:

Absolute neutrophil count (ANC) >1.5 × 10⁹/L Platelets >100 × 10⁹/L Hemoglobin >100 g/L Serum total bilirubin <1.5 × ULN ALT and AST <3 × ULN Creatinine clearance (CCr) >60 mL/min

* Voluntarily sign the informed consent form, able to understand and comply with study requirements.

Exclusion Criteria:

* Known allergy to any component of the study drugs.
* Prior treatment with any CTLA-4 targeting medication.
* Adverse reactions from previous anti-cancer therapy have not recovered to ≤ Grade 1 (per CTCAE v5.0) (except for toxicities without safety risk per investigator's judgment, e.g., alopecia).
* History of other malignancies within the past 5 years, except for cured malignancies.
* Severe comorbid conditions, including but not limited to:

Extensive interstitial lung disease requiring medication. Active or uncontrolled infections (e.g., tuberculosis, HIV). Decompensated liver disease, active hepatitis, or active bleeding. History of cerebrovascular accident or pulmonary embolism. Active, known, or suspected autoimmune diseases. Active infection requiring systemic anti-infective therapy.

* Ascites with depth >5 cm measured by ultrasound or CT, OR ascites causing severe symptoms (e.g., abdominal distension, dyspnea, circulatory dysfunction) significantly impacting physical function or study safety.
* Pregnant, planning pregnancy, or lactating women.
* Any other condition deemed by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult female patients (aged 18-75) with recurrent or metastatic cervical cancer whose disease has progressed after prior treatment with a PD-1 or PD-L1 inhibitor. Participants must have at least one measurable lesion, an ECOG performance status of 0 or 1, and adequate organ function.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment until disease progression, unacceptable toxicity, or any other discontinuation criterion is met (assessed approximately every 8 weeks for up to 24 months)
  The proportion of participants achieving a best overall response of Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Tumor assessments are performed by the investigators via computed tomography (CT) or magnetic resonance imaging (MRI) scans.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment until disease progression or death (assessed approximately every 8 weeks for up to 24 months).
  The time from the start of study treatment until the first documentation of disease progression as per RECIST 1.1, or death from any cause, whichever occurs first.
Duration of Response (DoR) | From the first recorded response until disease progression or death (assessed approximately every 8 weeks for up to 24 months).
  The time from the first documentation of objective response (CR or PR) per RECIST 1.1 until the first documentation of disease progression or death from any cause.
Disease Control Rate (DCR) | From enrollment until disease progression, unacceptable toxicity, or any other discontinuation criterion is met (assessed approximately every 8 weeks for up to 24 months).
  The proportion of participants who achieve a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST 1.1, maintained for at least 4 weeks.
Overall Survival (OS) | From enrollment until death from any cause (assessed every 12 weeks during follow-up for up to 24 months).
  The time from the start of study treatment until death from any cause.